CLINICAL TRIAL: NCT04258670
Title: Spontaneous Antigenemia in Loiasis, A Study of the Loiasis Antigens Responsible for Cross-reactivity in the Rapid Diagnostic Test for Lymphatic Filariasis
Brief Title: Spontaneous Antigenemia in Loiasis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Washington University School of Medicine (Other)
Collaborators: Doris Duke Charitable Foundation (Other); Centre for Research on Filariasis and other Tropical Diseases (Unknown)
Responsible Party: Sponsor
Other Study IDs: 201909003
Record Dates: First submitted 2020-02-03; First posted 2020-02-06 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Loiasis; Lymphatic Filariasis
Keywords: diagnostics; cross-reactivity
MeSH Terms: conditions — Loiasis; Elephantiasis, Filarial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Plasma Buffy coat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cross-reactive loiasis: This cohort will prospectively enroll 50 adults (age 18+) with cross-reactive antigenemia based on a positive filariasis test strip (FTS) and L. loa Mf counts >20,000 Mf/mL.
  Interventions: Other: No intervention
- non-cross-reactive loiasis: This cohort will prospectively enroll 10 adults (age 18+) with a negative filariasis test strip (FTS) and L. loa Mf counts >20,000 Mf/mL.

INTERVENTIONS:
Other: No intervention — Patients in these cohorts will not be given anti-filariasis therapies because these drugs are not approved for use in patients with high worm burdens (>20,000 Mf/mL)
  Groups: Cross-reactive loiasis

SUMMARY:
This prospective study will enroll and follow 60 loiasis patients with high worm burden to monitor the spontaneous release of filarial antigen in peripheral blood. This study will define the cross-reactive antigen profile of persons with spontaneous loiasis antigenemia, and determine whether it varies with time.

DETAILED DESCRIPTION:
Global efforts to eradicate lymphatic filariasis (LF) depend on rapid diagnostic tests (RDTs) that detect Wuchereria bancrofti circulating filarial antigen but these tests are unreliable in African nations where Loa loa is co-endemic because they yield false-positive results in some individuals with loiasis. The goals of this project are to define the cross-reactive antigen profile of persons with spontaneous antigenemia, how it varies over time, and to determine which L. loa antigens in cross-reactive sera best distinguish loiasis cross-reactivity from LF.

This prospective study will prospectively enroll 50 adults who presented with cross-reactive antigenemia at screening and 10 negative controls. Participants will followed for one year and tested every three months for persistence of antigenemia.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Loiasis Mf count > 20,000 Mf/mL
* Resident of study area
* No evidence of severe or systemic comorbidities
* Consent to storage of blood samples for future study

Exclusion Criteria:

* Subject plans to move from the study area during subsequent 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in the Okola health district (Lékié Division, Centre Region, Cameroon), situated about 40km northeast of Yaoundé, the political capital city of Cameroon. The Okola health district is highly endemic for loiasis. Participant will be recruited among those excluded from an Onchocerciasis study due to high Mf counts >20,000/mL.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-01-23 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
prevalence of specific cross-reactive L. loa antigens at baseline | 1 day
  Prevalence of filariasis test strip (FTS) positive individuals at screening. Cross-reactive proteins in plasma will be identified by mass-spectrometry to identify a cross-reactive biomarker

SECONDARY OUTCOMES:
Recurrence of cross-reactive antigenemia | quarterly for 1 year
  To determine if the same antigens are present at each follow up

CONTACTS AND LOCATIONS:
Overall Officials: Philip Budge, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Centre for Research on Filariasis and other Tropical Diseases (CRFilMT), Yaoundé, Cameroon

IPD SHARING:
Plan to Share IPD: Yes
The deidentified IPD for all primary and secondary outcomes will be made publicly available either as a supplementary file in a research publication and/or made publicly available in a data repository maintained by the Becker Biomedical Library at Washington University.
Time Frame: The data will be made available following publication. It will remain available indefinitely.
Access Criteria: The data will be made publicly available.